CLINICAL TRIAL: NCT06005987
Title: Effect of a Mobile Application on Blood Sugar Testing Compliance in Pregnant Women With Diabetes
Brief Title: Mobile App Logging for Diabetes in Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carolyn Zahler-Miller (Other)
Responsible Party: Sponsor-Investigator, Carolyn Zahler-Miller, Associate Professor, Augusta University
Organization: Augusta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1992519
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Type 2 Diabetes
Keywords: technology in medicine; mobile applications; blood glucose monitoring; diabetes in pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to two arms. First is traditional logging of blood glucoses with standard paper form in the clinic. The second arm will log their blood glucoses with the OneTouch Reveal smart phone application.
Who Masked: Outcomes Assessor
Masking Description: Cannot mask participant who needs to use the mobile application, or their care provider, or the investigator who will need to teach the patient how to use the application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile App arm (Experimental): Patient will input their daily blood glucose levels (fasting and 2 hours after breakfast, lunch and dinner) into the OneTouch Reveal app
  Interventions: Behavioral: OneTouch Reveal application
- Paper Log Arm (No Intervention): Patients will input their daily blood glucose levels onto paper logs which is the current process in the prenatal clinic.

INTERVENTIONS:
Behavioral: OneTouch Reveal application — Evaluate if compliance with glucose logging and percentage of in range glucoses changes with use of a mobile application instead of paper logging
  Arms: Mobile App arm

SUMMARY:
To determine the effect of using a mobile app versus paper logs on compliance and percentage in range blood sugars in monitoring blood sugar in pregnant women with diabetes.

DETAILED DESCRIPTION:
Women with type 2 and gestational diabetes have to keep strict logs of their blood sugar and record blood sugar values 4 times per day (fasting and 2 hours after every meal). This is often the first time they've had to keep such strict logs. Patients are provided with paper logs to record their blood sugars, however these can be lost or damaged and often they are not brought back to clinic. Mobile apps can be used to record blood sugar as well. This study will be comparing compliance with recording blood sugar values as prescribed with paper logs versus a mobile app. Subjects will be recruited from the Augusta University downtown location obstetric clinics.

Qualifying subjects must be at least 18 years of age with a verified intrauterine pregnancy of at least 12 weeks gestation and must have preexisting type 2 diabetes or gestational diabetes diagnosed by 1h glucose tolerance test (GTT) > 200mg/dL or 3h GTT with 2 or more abnormal values. Exclusion criteria includes patients with less than 2 weeks expected to be remaining in pregnancy, Preexisting use of a continuous glucose monitor (CGM) or application to track blood sugar readings, and type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Verified intrauterine pregnancy
* At least 12 weeks gestation
* Diagnosed with either type 2 diabetes mellitus or gestational diabetes mellitus.

Exclusion Criteria:

* Patients with less than 4 weeks anticipated to be remaining in pregnancy
* Pre-existing use of a continuous glucose monitor or other mobile application for glucose tracking
* Type 1 diabetes mellitus
* Non-English speaking patients

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must be pregnant.
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Compliance | 4 weeks
  percentage of actual blood glucose values logged compared to expected.

SECONDARY OUTCOMES:
Percentage of in-range blood glucose levels | 4 weeks
  Percentage of blood glucose levels in pregnancy appropriate range out of total blood glucose levels logged.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Keipper, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study completion and for 2 years afterwards
Access Criteria: contact study PI